CLINICAL TRIAL: NCT00003736
Title: Pilot Study: High Risk Breast Cancer Screening Pilot Study
Brief Title: MRI for Detecting Cancer in Women Who Are at High Risk of Developing Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Screening
Other Study IDs: CDR0000066851; UPCC-ACR-6884; UPCC -IBMC-6884
Record Dates: First submitted 1999-11-01; First posted 2003-08-20 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — motexafin gadolinium; Biopsy; Magnetic Resonance Spectroscopy

INTERVENTIONS:
Drug: motexafin gadolinium
Procedure: biopsy
Procedure: breast imaging study
Procedure: comparison of screening methods
Procedure: magnetic resonance imaging
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Screening tests may help doctors detect cancer cells early and plan more effective treatment for breast cancer. Diagnostic procedures such as MRI may improve the ability to detect breast cancer.

PURPOSE: Screening and diagnostic trial to study the effectiveness of MRI scans in women who are at high risk for developing breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Estimate the diagnostic yield and positive predictive value of breast magnetic resonance imaging (MRI) for the detection of cancer in women who are at greater than 25% lifetime risk for developing breast cancer.
* Compare the diagnostic yield and positive predictive value of MRI with conventional breast cancer screening (mammography and physical examination) for the detection of breast cancer in women with a greater than 25% lifetime risk of developing breast cancer.

OUTLINE: All patients receive a physical exam within 90 days of initial MRI scan. Patients undergo a two view screening mammogram within 3 months prior to study entry. Patients undergo an MRI with gadolinium contrast at entry. All lesions identified as suspicious on physical examination, mammography, or MRI undergo a core needle or excisional biopsy.

PROJECTED ACCRUAL: A total of 200 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients at greater than 25% lifetime risk for breast cancer on the basis of family history or a genetic test
* Prior breast cancer allowed if patient meets the greater than 25% lifetime risk

  * Patients with greater than 5 years since diagnosis must have at least 50% probability for developing breast cancer by the Couch model or be positive for BRCA1 or BRCA2 mutation
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 25 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No contraindications to MRI scan including patients with pacemakers, magnetic aneurysm clips or other implanted magnetic devices, or severe claustrophobia
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 25 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 1999-06; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Schnall, PhD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (12):
- United States (11):
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Roswell Park Cancer Institute, Buffalo, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Result] Lehman CD, Blume JD, Thickman D, Bluemke DA, Pisano E, Kuhl C, Julian TB, Hylton N, Weatherall P, O'loughlin M, Schnitt SJ, Gatsonis C, Schnall MD. Added cancer yield of MRI in screening the contralateral breast of women recently diagnosed with breast cancer: results from the International Breast Magnetic Resonance Consortium (IBMC) trial. J Surg Oncol. 2005 Oct 1;92(1):9-15; discussion 15-6. doi: 10.1002/jso.20350. PMID 16180217
- [Result] Lehman CD, Blume JD, Weatherall P, Thickman D, Hylton N, Warner E, Pisano E, Schnitt SJ, Gatsonis C, Schnall M, DeAngelis GA, Stomper P, Rosen EL, O'Loughlin M, Harms S, Bluemke DA; International Breast MRI Consortium Working Group. Screening women at high risk for breast cancer with mammography and magnetic resonance imaging. Cancer. 2005 May 1;103(9):1898-905. doi: 10.1002/cncr.20971. PMID 15800894